CLINICAL TRIAL: NCT03787004
Title: A Placebo-Controlled, Two-Part Study With Single Dose and Multiple Ascending Oral Dose to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of CNTX-6970 in Healthy Subjects
Brief Title: A Placebo-Controlled, Two-Part Study, Oral Dose to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of CNTX-6970 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNTX-6970-HV-102
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Chronic Pain; Nociceptive Pain
Keywords: Chronic Pain; Nociceptive Pain; Mixed Pain
MeSH Terms: conditions — Chronic Pain; Nociceptive Pain

STUDY DESIGN:
Masking Description: Part 1: Open Label Part 2: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Cohort 1 (Single Dose) (Experimental): Single 100 mg oral dose of CNTX-6970 (film-coated tablet or enteric-coated tablet)
  Interventions: Drug: CNTX-6970
- Part 1 Cohort 2 (Single Dose) (Experimental): Single 100 mg oral dose of CNTX-6970 film-coated tablet
  Interventions: Drug: CNTX-6970
- Part 2 (Multiple Ascending Dose) (Experimental): 100 mg, 300 mg, and 600 mg CNTX-6970 oral tablet
  Interventions: Drug: CNTX-6970
- Part 2 Placebo (Placebo Comparator): Placebo oral tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CNTX-6970 — Oral dose CNTX-6970
  Arms: Part 1 Cohort 1 (Single Dose); Part 1 Cohort 2 (Single Dose); Part 2 (Multiple Ascending Dose)
Other: Placebo — Oral dose placebo
  Arms: Part 2 Placebo

SUMMARY:
A Phase 1, placebo-controlled, two part study with either single dose or multiple increasing oral dose to evaluate the safety, pharmacokinetics, and pharmacodynamics of CNTX-6970 in healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Is in good general health as determined by the Investigator's review
* Has a body mass index (BMI) between 18 and 35kg/m^2, inclusive
* For females, is not currently pregnant or breastfeeding and is either of non-childbearing potential or willing to use an adequate method of birth control
* For males, must agree to use barrier contraception and not to donate sperm

Key Exclusion Criteria:

* Has a history of cardiac disease, including congestive heart failure, angina, or any arrhythmia
* Has diabetes mellitus, acromegaly, clinically active thyroid disease, or other active endocrinopathy
* Has any history or currently active type of cancer except excised or cured basal cell carcinoma
* Has a gastrointestinal disorder that could interfere with the absorption of orally administered drugs
* Has asthma or other severe respiratory disease (e.g., chronic obstructive pulmonary disease) requiring daily prescription medicine
* Currently has kidney, neurologic, metabolic, or liver disease, or other organ system disease
* Has a history, current evidence, or is being treated for depression, suicidal ideation, suicide attempt, or any other current psychiatric condition requiring active treatment
* Has an immunological disorder such as, but not limited to, human immunodeficiency virus (HIV), acquired, or congenital immune deficiency syndrome; autoimmune diseases, such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, seronegative spondyloarthropathies or vasculitis, or any infection
* Has positive screening test for hepatitis B virus (HBV) or hepatitis C virus (HCV);
* Is pregnant, lactating, or planning a pregnancy during the study
* Has used any prescribed medication within 30 days prior to the first admission or has plans to use any prescribed medication during the study (with the exception of hormonal contraceptives)
* Has used within 14 days prior to the first admission or has plans to use during the study any over-the-counter medicinal products, including herbal and dietary supplements (except for occasional use of acetaminophen or NSAIDs, such as ibuprofen or naproxen; calcium; or Vitamin D)
* Use of any of the following:

  * Human growth hormone, octreotide, anti-diabetic medication, or thyroid suppressors or supplements
  * Immunosuppressive drugs within 30 days of study start, or 5 half-lives of the drug (whichever is longer), or plans to use during the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
CNTX-6970 Pharmacokinetics - fasted state or high-fat standardized meal | Up to Day 3
  Food effects on pharmacokinetics of CTNX-6790 for Part 1 participants
CNTX-6970 Pharmacokinetics - AUC0-t | Up to Day 13
  Systemic exposure to CNTX-6970 measured by AUC0-t
CNTX-6970 Pharmacokinetics - AUC0-inf | Up to Day 13
  Systemic exposure to CNTX-6970 measured by AUC0-inf
CNTX-6970 Pharmacokinetics - Cmax | Up to Day 13
  Systemic exposure to CNTX-6970 measured by Cmax
CNTX-6970 Pharmacokinetics - tmax | Up to Day 13
  Systemic exposure to CNTX-6970 measured by tmax
CNTX-6970 Pharmacokinetics - t1/2 | Up to Day 13
  Systemic exposure to CNTX-6970 measured by t1/2

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) (safety and tolerability) | Up to Day 13
  Number of participants with TEAEs, which includes laboratory test variables
CNTX-6970 Pharmacodynamics - Emax | Up to Day 13
  Pharmacodynamic effect on MCP-1 and RANTES measured by Emax
CNTX-6970 Pharmacodynamics - PD tmax | Up to Day 13
  Time to maximum pharmacodynamic effect on MCP-1 and RANTES measured by tmax

CONTACTS AND LOCATIONS:
Overall Officials: Randall M. Stevens, MD, Study Chair — Centrexion Therapeutics
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States